CLINICAL TRIAL: NCT00010517
Title: Acupuncture in the Treatment of Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: R01 AT000001-01M; R01AT000001-01 (NIH); NCT00004534 (obsolete NCT alias)
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2008-03-07 (Estimated); Status verified 2008-03

CONDITIONS: Depressive Disorders; Depression
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — Acupuncture Therapy

INTERVENTIONS:
Procedure: Acupuncture

SUMMARY:
The current large randomized placebo-controlled trial is testing the ability of acupuncture to treat major depression. The study is unique in that treatment effects will be from the perspective of both Western psychiatry and Chinese medicine.

DETAILED DESCRIPTION:
Depression is an unfortunately common condition for which people often seek alternative (non-Western) treatments, perhaps because conventional treatments do not consistently provide lasting relief. A pilot study (Allen, Schnyer and Hitt, 1998) suggests that acupuncture, a popular but under-researched alternative treatment derived from Chinese medicine, holds sufficient promise as a treatment for depression to warrant a larger-scale clinical trial. The investigators propose to conduct a larger-scale test of the efficacy of acupuncture in this trial. Because relapse and recurrence of Major Depression are quite common, the investigators also will assess the clinical status of participants for 18 months after treatment concludes. In the first phase of this double-blind randomized clinical trial, 150 men and women meeting criteria for Major Depression will be randomly assigned to a treatment approach or to a waitlist control. All participants will ultimately receive acupuncture designed to address their own particular constellation of depressive symptoms. At the end of this first phase, blind assessments will be used to compare treatment effects from the perspectives of both Western psychiatry and Chinese medicine. After this treatment phase, participants will be assessed several times over the next 18 months. The study is designed to evaluate the efficacy and clinical significance of acupuncture as a treatment for Major Depression, and to examine the convergence of Western-based and Chinese-medicine-based outcome measures. Finally, the study will determine whether changes in energetic pattern mediate changes in Western defined depression severity, and explore whether patient and history variables predict responses to acupuncture treatments.

ELIGIBILITY:
Inclusion Criteria:

* Must meet criteria for Major Depression.
* Must be free of other mental or physical disorders that could cause depression, and also free from conditions that would typically exclude participants from trials involving pharmacologic antidepressants.
* Cannot be receiving other treatments or require immediate clinical attention.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1997-09; Study Completion 2002-04

CONTACTS AND LOCATIONS:
Overall Officials: John J. Allen, PhD, Principal Investigator — University of Arizona, Department of Psychology
Locations (1):
- University of Arizona, Tucson, Arizona, United States

REFERENCES:
- [Derived] Allen JJ, Schnyer RN, Chambers AS, Hitt SK, Moreno FA, Manber R. Acupuncture for depression: a randomized controlled trial. J Clin Psychiatry. 2006 Nov;67(11):1665-73. doi: 10.4088/jcp.v67n1101. PMID 17196044